CLINICAL TRIAL: NCT00289926
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, 52-week Study to Evaluate the Efficacy and Safety of Oral DHEA Therapy for Postmenopausal Women on Sexual Function, Wellbeing and Vasomotor Symptoms
Brief Title: Efficacy and Safety of Oral DHEA Therapy for Postmenopausal Women on Sexual Function, Wellbeing and Vasomotor Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Professor Susan Davis, Professor of Women's Health, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WHP 200501; NCT00394342 (obsolete NCT alias)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Quality of Life; Menopausal Syndrome; Libido Disorder
Keywords: low libido; lack of wellbeing
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dehydroepiandrosterone (Experimental): 50.0mg dehydroepiandrosterone capsule, by mouth, daily for 12 months
  Interventions: Drug: dehydroepiandrosterone
- Placebo (Placebo Comparator): Placebo capsule consists of 298.5 mg /capsule Microcrystalline Cellulose, NF 1.5 mg /capsule Magnesium Stearate, NF manufactured to mimic dehydroepiandrosterone capsule
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dehydroepiandrosterone — dehydroepiandrosterone capsules 50.0 mg /capsule DHEA 248.5 mg /capsule Microcrystalline Cellulose, NF 1.5 mg /capsule Magnesium Stearate, NF in a 60 mg Capsule
  Other Names: DHEA
  Arms: dehydroepiandrosterone
Drug: placebo — Placebo capsules of 298.5 mg /capsule Microcrystalline Cellulose, NF 1.5 mg /capsule Magnesium Stearate, NF in a 60 mg Capsule manufactured to mimic the active DHEA capsule
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of oral Dehydroepiandrosterone (DHEA) 50mg daily, for 12 months in naturally menopausal women with low libido who are not receiving systemic oestrogen or oestrogen- progestin therapy.

Efficacy measures for the present study are effects on sexual function, wellbeing and menopausal symptoms. Safety measures will include endometrial assessment by transvaginal ultrasound (TVU), vital signs, lipid profiles, general electrolytes, effects on glucose metabolism and reports of adverse events.

DETAILED DESCRIPTION:
Dehydroepiandrosterone (DHEA) and its sulphate (DHEAS) are the most abundant sex steroids in women. Dehydroepiandrosterone sulphate (DHEAS), a unique secretory product of the adrenal gland, and DHEA are converted at various sites in the body, such as the brain, bone and adipose tissue to estrogen or testosterone and their various by-products. DHEAS and DHEA levels decline with age and there has been considerable conjecture that this results in a loss of well-being and libido. DHEA is available as an over-the-counter nutritional supplement in the United States, and is being increasingly prescribed and formulated by compounding pharmacies across Australia. However, there is a paucity of data regarding the effects of oral DHEA on the well-being, sexual function and safety in women. Previous studies evaluating the effects of DHEA on either postmenopausal women or women with adrenal deficiency (Addison's disease) have produced conflicting results, with some studies finding benefit in terms of sexual function and well-being while other studies have found no benefit. Therefore, there is a need for an appropriately powered randomized controlled trial of the effects of DHEA therapy on sexual function and well-being in postmenopausal women. In addition, as DHEA may be metabolized to estrogens, whether DHEA will alleviate vasomotor symptoms merits evaluation. The effects of DHEA on the endometrial (uterine) lining requires assessment, given its potential to be converted to estrogen.

The primary aim of the current study will be to assess the effects of DHEA therapy in naturally menopausal women on sexual function using the Sabbatsberg Self-Rating Scale (SSS) over 12 months in a randomized placebo controlled trial. In addition the effects on well-being will be assessed by the Psychological General Well-Being (PGWB) Index and menopausal symptoms will be evaluated by the Menopause Quality of Life (MENQOL) Intervention Questionnaire. A diary record will also be employed to assess the effects on sexual function. Safety will be assessed over the entire study. Participants will also undergo a transvaginal ultrasound (TVU) at the beginning and end of the study, to determine whether DHEA affects the endometrial lining.

This randomized, double-blind, placebo-controlled study will be conducted in 240 women over a 52-week period. Women will be randomized to receive either placebo or DHEA (50 mg/day) for a 52-week period. It is anticipated that the study will require a 6-month recruitment period. The study duration will be approximately 56 weeks, with a 4-week screening period and treatment period of 52 weeks. The study will be conducted over approximately 13 months. This is a single-centre study and will be conducted at the Alfred Hospital.

Potential participants will be generally healthy women aged 40 - 65 years who have undergone a natural menopause and are in a stable monogamous sexual relationship and not using hormone therapy (HT).

Participants are required to attend 6 clinic visits over a blinded treatment period of 52 weeks. Informed consent will be obtained from the participant prior to the commencement of any study procedure at the first clinic visit. If participants are eligible, they will be asked to return at the end of the screening period to be randomized and commence treatment. During the treatment period, participants will take one capsule daily (placebo or DHEA 50 mg). All participants will return to the clinic 5 more times, at weeks 0, 12, 26, 38 and 52 for assessments of efficacy and safety. Blood tests will be collected at Weeks -4, 0, 12, 26 and 52 to assess safety and hormone levels. Prior to commencing the study, participants will require a mammogram if this has not been done within 12 months of study entry. A transvaginal ultrasound will be performed to assess endometrial thickness prior to commencement of the trial. A Papanicolaou smear will also be performed if the cervix is still present, in those women where a Pap smear has not been done within 12 months of screening. These investigations, except the mammogram and Pap smear, will be repeated at the completion of the study. All participants will have a complete physical examination which will include an assessment of vital signs, breast examination, and internal and external pelvic examination to assess for clitoromegaly (clitoral enlargement). Skin evaluations for scalp hair loss, hirsutism and acne, and assessment for voice changes will be made throughout the study. Participants will be required to complete various questionnaires to assess sexual function (SSS), menopausal symptoms (MENQUOL Intervention) and general well-being (PGWB) at Weeks 0, 12, 26 and 52. Participants will also record satisfactory sexual events in a 28 day diary which will be done in the 4 weeks prior to Weeks 0, 12, 26 and 52.

ELIGIBILITY:
Inclusion Criteria:

Women who:

1. are 40 to 65 years of age, at least 12 months postmenopausal (no spontaneous menses in the last 12 months, or be over the age of 55 years, or hysterectomy with one or both ovaries in situ and follicle-stimulating hormone [FSH] > 20 IU/L. (An FSH > 20 IU/L will also be used to confirm menopausal status in non-hysterectomised women < 55 years, where menopausal status is unclear.)
2. are sexually active -defined as being involved in any form of sexual activity at least once a month. Women do not require a partner.
3. have a body mass index (BMI) 18-34 kg/m2.
4. answer affirmatively to the following questions:

   * In previous years did you find sexual activity satisfying?
   * Do you feel that you have experienced a significant decrease in your desire or interest?
   * Would you like an improvement in your desire or interest for sexual activity?
   * Would you like to be treated for this?
5. Have a clinically acceptable screening bilateral mammogram
6. Have ≤ 4 mm endometrial double thickness and no other abnormal findings on TVU if not hysterectomised.
7. Have a clinically acceptable Pap smear if the cervix is present,
8. Be able and willing to participate in the study as evidenced by providing written informed consent.
9. have a baseline DHEAS level of < 2.1 umol/L

Exclusion Criteria:

1. Have a BMI < 18 or > 34 kg/m2
2. Dyspareunia not alleviated by use of lubricants.
3. Severe depression (Beck Depression Inventory Score-II [BDI] > 20).
4. Have partnership problems. This will be established by interview by asking the following questions if a woman is in a specific relationship:

   1. Are you satisfied with your partner as a friend?
   2. Do you have concerns about your relationship?
5. Have used recent androgen therapy (testosterone implant within the last 28 weeks, transdermal testosterone cream within the last 8 weeks, tibolone within the last 12 weeks, oral testosterone within the last 4 weeks and injected testosterone within the last 6 weeks).
6. Have used treatment for depression (antidepressants, antipsychotics, antiepileptics) within 2 months ).
7. Have known severe psychiatric illness.
8. Have used estrogen, including vaginal conjugated equine estrogen, vaginal ring delivering up to 7.5 µg/day, or estrogen-progestin combinations in the last 2 months. (Use of Ovestin or Vagifem pessaries or cream will be allowed.)
9. Used phytoestrogens within 1 week prior to Week -4 (Visit 1). (Women will be allowed to participate in this trial, provided they cease using phytoestrogens for at least 1 week before visit 1.)
10. Have renal disease, liver disease, epilepsy, or diabetes mellitus or any other major illness that has occurred within the last 6 months.
11. Therapies known to induce liver enzyme metabolism or alter the metabolism of DHEA e.g. antiepileptics, dexamethasone, or antituberculous drugs.
12. Undiagnosed genital bleeding.
13. Have moderate to severe acne or hirsutism, have used antiandrogen therapy for acne or hirsutism in the preceding 5 years, or have androgenic alopecia.
14. Active malignancy or treatment for malignancy in the preceding 5 years (excluding non-melanotic skin cancer).
15. Report alcohol consumption > 3 standard drinks per day.
16. Have a history of cerebrovascular disease, thromboembolic disorders, myocardial infarction or angina at anytime before study entry or thrombophlebitis within the last 5 years.

16. An abnormal thyroid-stimulating hormone (TSH) value at screening (however, participants with an abnormal TSH, but normal free T4 and free T3 and no clinical signs or symptoms of thyroid disease, with or without replacement treatment, may be admitted to the study).

17. Have abnormal liver function (LFTs) which is significant and/or an ALT or AST > 3 times the upper limit of normal or bilirubin > 2 times the upper limit of normal.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The assessment of the efficacy of oral DHEA therapy in postmenopausal women on sexual function | 6 months

SECONDARY OUTCOMES:
Safety of DHEA treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Davis, MBBS, PhD, Principal Investigator — Monash University
Locations (1):
- Women's Health Research Program, Monash University, The Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Women's Health research Program — http://womenshealth.med.monash.edu.au